CLINICAL TRIAL: NCT02934984
Title: Analysis of Factors Related to Pancreatic Cancer Recurrence Using Circulating Cell-free Tumor DNA(ctDNA)
Brief Title: Circulating Cell-free Tumor DNA(ctDNA) in Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JooKyung Park, Clinical assistant professor, Samsung Medical Center
Other Study IDs: 2016-07-054
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; recurrence; DNA
MeSH Terms: conditions — Pancreatic Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigator will collect peripheral blood cell-free tumor DNA(ctDNA) in pancreatic cancer patients, benign pancreas disease patients and healthy population.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the study is to evaluate whether peripheral circulating cell-free tumor DNA(ctDNA) can help early screening of pancreatic cancer recurrence or not. And we are also planning to evaluate correlation between ctDNA with clinical outcome of pancreatic cancer.

DETAILED DESCRIPTION:
In the formation and growth of a primary tumor, cells can released into the bloodstream. There are many researches for these circulating tumor cells(CTC) And recently circulating cell-free tumor DNA(ctDNA) released from apoptotic or necrotic tumor cells has developed. At one report which checked ctDNA level after operation of colon cancer patients, they suggested that ctDNA could show recurrence of cancer several months earlier than the conventional follow up imaging. And several reports suggested that ctDNA can invade host cell and change host cell biology, which can evoke cancer metastasis.

So in this study, the investigator will collect ctDNA of pancreatic cancer patients, benign pancreatic disease patients, and healthy population. And the investigator will evaluate whether peripheral ctDNA can help early screening of cancer recurrence. And we will study about genomic signature of ctDNA to evaluate relationship between ctDNA and clinical outcome of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Comparative group : Pancreatic cancer patients who progress endoscopic ultrasonography fine-needle aspiration (EUS-FNA) for pancreatic cancer diagnosis, pancreatic cancer patients who are in operable stage
* Control group : Benign pancreas disease patients who progress EUS-FNA for diagnosis, healthy population

Exclusion Criteria:

* Foreigners
* Pancreatic cancer patients who have other cancer
* Patients who impossible to consent to study by own

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive pancreatic cancer patients who received EUS-FNA for diangosis and undergo operation, benign pancreas disease patients who received EUS-FNA for diagnosis, healthy population
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2020-07 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Rates of recurrence in pancreatic cancer patients | 36 months

SECONDARY OUTCOMES:
Rates of death in pancreatic cancer patients | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided